CLINICAL TRIAL: NCT06954662
Title: Comparison of Whey Protein and Amino Acid Supplementation on Amino Acid and Levodopa Concentrations in People With Parkinson's Disease
Brief Title: A Targeted Amino Acid Supplement for People With Parkinson's Disease
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Cristina Colón-Semenza, Assistant Professor, UConn Health
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 24-017S-1
Record Dates: First submitted 2025-03-28; First posted 2025-05-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease, Idiopathic
Keywords: Nutrition; Amino acid supplementation; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a prospective, double-blind, randomized control trial with a repeated measures design in a single group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Whey Protein Supplement (WP-S) (Active Comparator): Whey protein is one of the primary proteins found in all dairy products. It is a complete protein as it contains all the essential amino acids. It is commercially available as a dietary supplement (a standard 20 g dose of whey).
  Interventions: Dietary Supplement: Whey Protein Supplement
- Isonitrogenous Placebo Supplement (CON-S) (Placebo Comparator): The control supplement used in this study is an isonitrogenous placebo beverage. This supplement will consist of an inert amino acid (alanine) with the same amino acid load as the WP-S and AA-S (16.2 g).
  Interventions: Dietary Supplement: Isonitrogenous Placebo Supplement
- Amino acid supplement (AA-S) (Experimental): designed off the amino acid composition of the why protein supplement, but then was modified to minimize interference with levodopa by reducing the quantity of amino acids which are known to interfere with levodopa, which collectively resulted in a 59% reduction in competing amino acids. Additionally, the concentrations of other non-competing amino acids were modified in order to fill the previously identified nutritional deficiency observed in people with PD.
  Interventions: Drug: Amino acid supplement

INTERVENTIONS:
Drug: Amino acid supplement — a targeted amino acid supplement designed to provide dietary nutrients that are commonly deficient in people with PD while minimizing interference with L-Dopa medication
  Other Names: AA-S
  Arms: Amino acid supplement (AA-S)
Dietary Supplement: Whey Protein Supplement — Whey protein is one of the primary proteins found in all dairy products. It is a complete protein as it contains all the essential amino acids. We will use a 20 gram dose.
  Other Names: WP-S
  Arms: Whey Protein Supplement (WP-S)
Dietary Supplement: Isonitrogenous Placebo Supplement — The control supplement used in this study is an isonitrogenous placebo beverage. This supplement will consist of an inert amino acid (alanine) with the same amino acid load as the whey protein and the targeted amino acid supplement (16.2 grams).
  Other Names: CON-S
  Arms: Isonitrogenous Placebo Supplement (CON-S)

SUMMARY:
The goal of this clinical trial is to learn if an amino acid supplement that is specifically made for people with Parkinson disease can improve nutrition without interfering with dopamine medication in people living with Parkinson disease. The main question it aims to answer is:

• Does an amino acid supplement that is specifically made for people with Parkinson disease have short-term improvements in nutrition deficiencies, while minimally interfering with Parkinson disease medication?

Researchers will compare the short-term effects of this specialized nutrition supplement to a supplement that is available for everyone to purchase in a store (whey protein supplement-a milk by-product) and to an inactive supplement. Researchers will then check for the indicators of nutrition levels and the presence of dopamine medication in the blood. Researchers will also assess mood and movement abilities in participants.

Participants will be asked to:

* attend 4 study visits over the course of 4 weeks (initial orientation visit plus 3 intervention visits).
* drink one of the 3 supplements (supplements will be mixed into water to create a beverage) at each of the 3 intervention visits.

  * participate in blood drawings and mood and movement assessments at each of the intervention visits.
  * engage in a phone call after each intervention visit to determine any delayed responses.

DETAILED DESCRIPTION:
This is a prospective, double-blind, randomized control trial with a repeated measures design. After being screened via phone screens and completing an initial visit that includes additional in person screening and the collection of descriptive information, participants will be invited to take part in three experimental sessions. On three separate days participants with idiopathic Parkinson's Disease and taking a stable dose of dopamine replacement medication, 2-3 hours after a standardized low-protein meal, will orally take a habitual dose of L-Dopa medication and then engage in one of the three interventions 1) WP-S: whey protein supplement (20 g), 2) AA-S: targeted amino acid supplement (equivalent amino acid load to whey protein beverage) 3) CON-S: an isonitrogenous placebo beverage (equivalent amino acid load to whey protein beverage), prescribed in a randomized and counterbalanced manner. Prior to, and up to 3 hours after medication, blood samples will be collected every 15 min for 90 min and every 30 min thereafter and then analyzed to determine circulating L-dopa and amino acid profiles using high-performance liquid chromatography. During this observation period changes in both motor (Movement Disorder Society-Unified Parkinson's Disease Rating Scale Part 3 (MDSUPDRS III), finger tapping, and Timed Up and Go Test) and non-motor disease symptoms (Profile of Mood State with component analysis of depression, fatigue, and anxiety) will be measured every 30 minutes.

All supplements will be provided for the study in coded prepackaged envelopes by an independent nutritional supplement company based on the formulas provided below, to ensure double blinding.

Whey Protein Supplement (WP-S): Whey protein is one of the primary proteins found in all dairy products. It is a complete protein as it contains all the essential amino acids. A previous investigation has been performed looking at the long -term (6 months) effects of whey protein supplementation on health and disease symptoms of people with Parkinson's Disease. This study validated the safety and efficacy of whey protein supplementation in people with Parkinson's Disease, but a non-significant increase in disease symptoms (during medication off time) was reported. Similar to this previous study, we will use a standard 20 g dose of whey protein.

Targeted Amino Acid Supplement (AA-S): Previous studies have investigated the long-term (6 months) effects of amino acid supplementation on health and disease symptoms of people with Parkinson's Disease. The previous whey protein study, and the previous amino acid supplement study, validated the safety and efficacy of an amino acid supplement in people with Parkinson's Disease but a non-significant increase in disease symptoms (during medication off time) was reported. However, the supplement in these studies was not designed to minimize the components which could interfere with levodopa medication.

In contrast, the AA-S used in the present study was designed off the amino acid composition of WP-S, but then was modified to minimize interference with levodopa by reducing the quantity of amino acids which are known to interfere with levodopa (large neutral amino acids), which collectively resulted in a 59% reduction in competing amino acids. Additionally, the concentrations of other non-competing amino acids were modified in order to fill the previously identified nutritional deficiency observed in people with PD.

Isonitrogenous Placebo Supplement (CON-S): The control supplement used in this study is an isonitrogenous placebo beverage. This supplement will consist of an inert amino acid (alanine) with the same amino acid load as the WP-S and AA-S (16.2 g).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic Parkinson disease by patient report
* 55 years or older
* Has been using dopamine replacement medication (e.g. levodopa) for at least 2 years.
* On a stable dose of dopamine replacement medication for at least 3 months with no plans for change in the next two months.

Exclusion Criteria:

* Apparent cognitive impairment as determined by phone screening (TICS)
* Diagnosis of Parkinsonism or atypical Parkinson's Disease
* Are prescribed a dopamine antagonist
* Any unstable medical condition
* Any known bleeding disorder or currently taking blood thinners
* Using deep brain stimulation
* Gastric or bowel resection surgery

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Circulating levodopa | study session 2 (Week 2), 3 (Week 3), and 4 (Week 4). Each session will last approximately 3-4 hours.
  Circulating levodopa will be measured from the 10 blood samples at each of the three study visits.
Circulating amino acids concentrations | Session 2 (Week 2), Session 3 (Week 3), Session 4 (Week 4)
  High performance liquid chromatography will be used to assess amino acid concentrations in blood samples (10) from each intervention session

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale, Part III | This test will be performed prior to medication (Pre/+0 minutes) and at the end of testing (+180 minutes) at each of the 3 intervention sessions (Session 2/Week 2, Session 3/Week 3, Session 4/Week 4)
  Disease motor symptoms will be assessed via Part 3 of the UPDRS. Research staff that have completed training to administer and grade this test by the International Parkinson and Movement Disorder Society will complete this assessment. This portion of the UPDRS is designed to test motor symptoms related to Parkinson's Disease. The test includes quick clinical assessments of passive rigidity, finger and toe tapping, hand and forearm movement, chair standing, gait (10 meter) assessment, and postural assessment.
Timed Up and Go Test | This test will be performed every 30 minutes (+0, +30, +60, +90, +120, +150, and +180 minutes) at each of the intervention sessions (Session 2/Week 2, Session 3/Week 3, Session 4/Week 4).
  The timed up and go test will be performed as an additional physical symptom assessment. In this test the participant will start in a seated position, then stand up, walk 3 meters and then turn around and return to the chair.
Abbreviated Profile of Mood State | This test will be performed prior to medication (Pre/+0 minutes) and at the end of testing (+180 minutes) at each intervention session.
  Abbreviated Profile of Mood States (POMS) Questionnaire: This an assessment of current mood state. It is a 40-item self-report survey that evaluates the degree to which a participant is feeling a selected emotion at the moment.
30 second Finger Tapping | This test will be performed every 30 minutes (+0, +30, +60, +90, +120, +150, and +180 minutes) at each intervention session
  The 30 second finger tapping test is an assessment of fine motor control. The participant will sit upright in a chair with their most affected (with the greatest disease symptoms) hand positioned over a tablet. In this position the participant will tap the screen as many times as they can for 30 seconds, and the total number of taps will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Colon-Semenza, PT, MPT, PhD, Principal Investigator — University of Connecticut; Jacob Earp, PhD, Principal Investigator — University of Connecticut
Locations (1):
- UConn Health, Clinical Research Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
The funding for reviewing requests, storing and managing data, and sharing IPD is undetermined at this time.

REFERENCES:
- [Background] Earp JE, Colon-Semenza C, LoBuono DL. Considerations for developing a targeted amino acid supplement for people with Parkinson's disease that promotes health while accounting for pathophysiology and medication interference. Nutr Rev. 2023 Jul 10;81(8):1063-1076. doi: 10.1093/nutrit/nuad008. PMID 36809398